CLINICAL TRIAL: NCT00622817
Title: Double Blinded Controled Study:Treatment With Adrenaline Inhalation Versus Nasal Decongestant Drops for Bronchiolitis
Brief Title: The Influence of Inhaled Adrenalin Versus Decongestant as a Local Nasal Treatment in Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Schneider Children's Medical Center, Israel, Sackler Medical Center, tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2848
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2002-02

CONDITIONS: Bronchiolitis
Keywords: Epinephrine; Nasal decongestant; RSV; xylometazoline; Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients are treated with inhalation of epinephrine 1mg and nasal drops of 0.9% saline for each nostril every twelve hours.
  Interventions: Drug: Epinephrine 1mg
- 2 (Experimental): Receive four inhalation of 0.9% saline four times a day and one nasal drop of xylometazoline HCL 0.05% to each nostril twice a day.
  Interventions: Drug: xylometazoline HCL 0.05%

INTERVENTIONS:
Drug: xylometazoline HCL 0.05% — Receive four inhalation of 0.9% saline four times a day and one nasal drop of xylometazoline HCL 0.05% to each nostril twice a day.
  Other Names: xylometazoline HCL = Otrivin nasal drops
  Arms: 2
Drug: Epinephrine 1mg — Patients are treated with inhalation of epinephrine 1mg and nasal drops of 0.9% saline for each nostril every twelve hours.
  Arms: 1

SUMMARY:
This was a randomized, double blinded, controlled trial. The aim of the study was to compare xylometazoline HCL nasal drops to inhalation of epinephrine as a treatment for bronchiolitis.

The study hypothesis is:xylometazoline HCL nasal drops treatment is good as epinephrine inhalation for treatment of bronchiolitis.

Signed informed consent was obtained from a parent of each child. And the human ethics committee of our hospital approved the study according to the principles of the Declaration of Helsinki.(Approved - 2002)

Patients:

65 infants who were admitted to Pediatric A- a general pediatric ward, in Schneider Children's Medical Center because of bronchiolitis during winter in two consecutive years 2004-2005.

The inclusion criteria were: Full term previously healthy Infants, ages 1-12 months, after informed consent was signed with clinical presentation of mild to moderate bronchiolitis according to a clinical score .Exclusion criteria were as follows: prematurity, congenital lung or cardiac disease, infants who had past hospitalization due to respiratory illness and severe bronchiolitis (score>7 with a range scale 0-10).

DETAILED DESCRIPTION:
All eligible patients were randomly assigned to one of two groups: Group 1 (control) received inhalation of epinephrine 1mg, in 2cc of 0.9% saline solution four times a day, and nasal drops of 0.9% saline for each nostril every twelve hours. Group 2 - the study group received four inhalation of 0.9% saline four times a day and one nasal drop of xylometazoline HCL to each nostril twice a day. This treatment continued until the patient was ready for discharge.

Patients were examined and evaluated at the study entry and were re-evaluated every 10-12 hours. Length of hospital stay,time to improve Oxygen saturation, time to the need of IV fluid and clinical score between the two groups of treatment were compared.

ELIGIBILITY:
Inclusion Criteria:

* Full term previously healthy Infants
* Ages 1-12 months
* After informed consent was signed with clinical presentation of mild to moderate bronchiolitis

Exclusion Criteria:

* Prematurity, congenital lung or cardiac disease
* Infants who had past hospitalization due to respiratory illness and severe bronchiolitis (score >7 with a range scale 0-10)

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2004-10; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Two years

SECONDARY OUTCOMES:
Time to improve oxygen saturation, comparison of clinical scores , Needs of IV fluids | 2 years

REFERENCES:
- [Derived] Livni G, Rachmel A, Marom D, Yaari A, Tirosh N, Ashkenazi S. A randomized, double-blind study examining the comparative efficacies and safety of inhaled epinephrine and nasal decongestant in hospitalized infants with acute bronchiolitis. Pediatr Infect Dis J. 2010 Jan;29(1):71-3. doi: 10.1097/INF.0b013e3181b0602e. PMID 19907355